CLINICAL TRIAL: NCT02177604
Title: Can Brief High-intensity Interval Training Mitigate the Adverse Consequences of High-fat Overfeeding?
Acronym: GAINHIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Adelaide (Other)
Collaborators: Royal Adelaide Hospital (Other); University of South Australia (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, Associate Professor, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140319
Record Dates: First submitted 2014-06-19; First posted 2014-06-27 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wingate HIT (Experimental): 7 days of high-fat overfeeding (50% excess calories) in conjunction 3 supervised sessions of Wingate High-intensity Interval Training.
  Interventions: Other: Wingate HIT; Other: High-fat overfeeding
- Modified HIT (Experimental): 7 days of high-fat overfeeding (50% excess calories) in conjunction with 3 supervised sessions of Modified High-Intensity Interval Training
  Interventions: Other: Modified HIT; Other: High-fat overfeeding
- No Exercise Control (Active Comparator): 7 days of high-fat overfeeding (50% excess calories) with no supervised exercise
  Interventions: Other: High-fat overfeeding

INTERVENTIONS:
Other: Wingate HIT — 3 sessions of Wingate based High-Intensity Interval Training (6-8 x 15 second "all out" sprints on a cycle ergometer interspersed by 2 minutes recovery)
  Arms: Wingate HIT
Other: Modified HIT — 3 sessions of Modified High-Intensity Interval Training (8 x 60 second sprints at approximately 90-95% VO2 peak on a cycle ergometer interspersed by 60 seconds recovery)
  Arms: Modified HIT
Other: High-fat overfeeding — 7 days of high-fat overfeeding (50% excess calories)

SUMMARY:
Previous research has shown that indulging in 50% more calories than required for as little as 3 days can significantly impact markers of metabolic health in lean and overweight individuals. Here, the investigators will determine if 3 brief sessions of high-intensity interval training can mitigate the adverse consequences of 7 days high-fat overfeeding in sedentary, overweight males.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (no more than 2 sessions of structured moderate intensity aerobic exercise or resistance training per week)
* Overweight (BMI 25-29.9 kg/m2)

Exclusion Criteria:

* Personal history of any major illness (i.e. cardiovascular disease, diabetes, hypertension, cancer, renal/liver impairments, major psychiatric disorders, eating disorders etc.)
* History of chest pain (either at rest or during exercise.)
* Abnormal resting ECG at screening visit
* Chronic use of any prescribed or non-prescribed medications (i.e. anti-hypertensive, statins, metformin, anti-inflammatories, antidepressants etc.)
* Blood pressure or blood lipids outside of reference ranges
* Serum ferritin <30ng/mL
* Uncontrolled asthma, current fever, or upper respiratory infection
* Current intake of > 140g alcohol/week
* Current smokers of cigarettes/cigars/marijuana
* Current intake of any illicit substance
* Experience claustrophobia in confined spaces
* Donated blood in the past 3 months
* Migraines
* Unable to comprehend study protocol
* Unable to perform exercise on a cycle ergometer at second screening visit

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in glucose metabolism | 1 week
  Changes in insulin and glucose area under the curve assessed via 75g Oral Glucose Tolerance Test.

SECONDARY OUTCOMES:
Change in plasma levels of cytokines | 1 week
  Change in plasma levels of adiponectin, irisin, sex hormone-binding globulin and c-reactive protein

OTHER OUTCOMES:
Change in mitochondrial metabolism | 1 week
  Changes in citrate synthase activity, mitochondrial DNA content and protein levels of PGC-1a
Change in resting energy expenditure | 1 week
  Changes in resting energy expenditure measured by metabolic cart
Change in cognitive function | 1 week
  Changes in cognitive function, assessed by a series of computer tasks involving vigilant attention and speed processing.

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Heilbronn, PhD, Principal Investigator — University of Adelaide
Locations (1):
- South Australian Health & Medical Research Institute, Adelaide, South Australia, Australia